CLINICAL TRIAL: NCT05818566
Title: The Challenge of Treating Orphan Diseases With Novel Therapies: Experience From One Adult Metabolic Clinic in Switzerland
Brief Title: Orphan Drugs for Inherited Metabolic Diseases
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Christel Tran, Principal investigator, University of Lausanne
Other Study IDs: 2022-01470
Record Dates: First submitted 2023-04-04; First posted 2023-04-19 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2023-11

CONDITIONS: Inborn Errors of Metabolism
Keywords: Orphan Drugs; Inherited Metabolic Diseases
MeSH Terms: conditions — Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to report and describe all the patients with confirmed diagnosis of inherited metabolic disease (IMD) treated with orphan medicinal products (OMPs) in a cohort of adult patients followed in a reference center for rare diseases (Lausanne University Hospital, CHUV) from 2017-2022.

DETAILED DESCRIPTION:
The development of novel therapies for inherited metabolic diseases, considered has OMPs, has improved the care of these patients. OMPs include a wide range of therapies from dietary products, enzyme replacement, substrate inhibitors, coenzyme replacement to more recently, gene therapy. Despite an increasing use of these therapies, they are still considered highly specialized treatments for very small groups of patients and share the characteristic of aiming to treat small populations with targeted therapies, which leads to higher costs and difficulties in obtaining clinical evidence. Drugs are approved for marketing and orphan designation by medical agencies based on their efficacy and safety.

In Switzerland, a separate country-specific process decides whether an approved drug is reimbursed. Because of the growing number of expensive OMPs, their reimbursement through public health insurances is increasingly manifesting itself as a moral dilemma for decision-makers. It may take a median of several years after submission of the first application by a pharmaceutical company for an orphan drug to become available to patients.

Considering the increasing number of OMP approvals and the still ethical challenge concerning their reimbursement, this study aims to share the experience of a single center in treating adult IMDs with OMPs but also in implementing novel therapies for rare diseases not yet covered by health insurers in Switzerland.

A database was created in 2017 including all patients with IMD followed at the Adult Metabolic Clinic in the CHUV. This database was part of a protocol submitted and approved by the Ethics committee (# 2017-02328). The results of this first analysis were published in the Journal of Orphan Rare Diseases. Investigators will use this database to identify all the patients treated with OMPs. Electronic and paper patient charts from the Division of Genetic Medicine will be reviewed for type of IMD and treatment. All variables will be entered in an excel database.

ELIGIBILITY:
Inclusion Criteria:

* Age = or > 16 years
* Biological and/or genetically confirmed diagnosis of IMD

Exclusion Criteria:

* Age < 16 years
* Document attesting refusal to participate

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient clinic for Adult patients with IMD from the Lausanne University Hospital (Division of Genetic Medicine)
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Specific diagnosis of Inherited Metabolic Diseases listed by their frequency | Day1
  Clinical outcome
Age at diagnosis (years/months) | Day1
  Clinical outcome
Current age (years/months) | Day1
  Clinical outcome
Specific treatment for inherited metabolic diseases | 5 years
  Treatment specific to each diseases including only OMPs

SECONDARY OUTCOMES:
Gender (Male/Female) | Day 1
  Demography outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Gariani K, Nascimento M, Superti-Furga A, Tran C. Clouds over IMD? Perspectives for inherited metabolic diseases in adults from a retrospective cohort study in two Swiss adult metabolic clinics. Orphanet J Rare Dis. 2020 Aug 18;15(1):210. doi: 10.1186/s13023-020-01471-z. PMID 32811506